CLINICAL TRIAL: NCT00533559
Title: Mechanism of Fatty Acid-induced Impairment of Glucose-stimulated Insulin Secretion - Effect of Buphenyl
Brief Title: Mechanism of Fatty Acid-induced Impairment of Glucose-simulated Insulin Secretion - Effect of Buphenyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Gary Lewis, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 07-0274-B; Canadian Diabetes Association (Other Grant/Funding Number: 777508221)
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes; Insulin Resistance
Keywords: type 2 diabetes; free fatty acids; insulin resistance; beta cell lipotoxic effect
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- buphenyl (Experimental)
  Interventions: Drug: sodium phenylbutyrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sodium phenylbutyrate — buphenyl, 7.5 gm/day for two weeks for two studies, one with saline and one admission with intralipid and heparin
  Arms: buphenyl
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
An increase of plasma free fatty acids impairs insulin secretion and insulin sensitivity, thereby playing an important role in causing type 2 diabetes. Lipotoxicity plays an important role in the progression from normal glucose tolerance to fasting hyperglycemia and coversion to frank type 2 diabetes. A recent publication in the journal Science showed that buphenyl, when given to obese diabetic mice, resulted in normalization of hyperglycemia, restoration of systemic insulin sensitivity, resolution of fatty liver disease and inhancement of insulin action in liver, muscle and adipose tissue. the mechanism of action is believed to be due to reduction of endoplasmic reticulum (ER) stress. Buphenyl is currently approved for the treatment of rare inherited disorders of the urea cycle. We plan to administer Buphenyl orally to humans at a dose far lower than that used for the treatment of urea cycle disorders for 2 weeks prior to the testing of pancreatic function. One potential mechanism whereby chromically elevated plasma FFAs and glucose impairment beta cell function and insuln sensitivity is by ER stress and this can be prevented by administeration of buphenyl.

DETAILED DESCRIPTION:
Each subject will undergo 4 studies, 4 weeks apart. Each study will consist of a 2 week treatment period with either Buphenyl or placebo, followed by 48 hour hospital stay to test insulin sensitivity and insulin secretion. The four studies are as follows: 1. 2-week placebo tablets followed by in hospital 48-hour infusion of normal saline prior to testing of insulin secretion and insulin sensitivity (CONTROL study), 2. 2-week placebo treatment followed by 48 hour infusion of intralipid and heparin to raise plasma free fatty acids 2-fold prior to testing of insulin secretion and insulin sensitivity (PLACEBO-INTRALIPID+HEPARIN study), 3. 2-week Buphenyl treatment followed by 48-hr infusion of intralipid and heparin to raise plasma free fatty acids 2-fold prior to testing of insulin secretion and insulin sensitivity (BUPOHENYL+INTRALIPID+HEPARIN study), 4. 2-week Buphenyl treatment followed by 48-hr infusion of normal saline prior to testing of insulin secretion and insulin sensitivity (BUPHENYL+SALINE study).

For two weeks prior to each admission to hospital and during each hospital admission subjects will ingest 5 tablets 3 times per day with meals (total of 15 tablets per day). For two of the 4 studies the tablet will contain Buphenyl (total of 15 tablets per day, each tablet of Buphenyl contains 500mg, total 7.5grams per day), whereas for the other two studies the tablet will be a placebo, containing no active ingredient. The study will be conducted as a single blind study, with the subject not knowing whether they are receiving a placebo or biphenyl. For safety reasons and since it will not influence the results of this study it will not be conducted as a double blind study. On each of four occasions, 4 weeks apart, after taking the tablets for 2 weeks, the subject will fast overnight for 12-hours prior to their admission to the Toronto General Hospital metabolic research ward for 48 hours to undergo testing as follows.

On the morning they are admitted an intravenous (iv) line will be placed in a superficial vein (under the skin) of each forearm (2 iv's, one iv in each arm). These intravenous lines will be used for blood sampling at regular intervals throughout the study and to infuse solutions. Blood samples will be drawn painlessly through the IV at timed intervals for the first two days. The total amount of blood to be taken for each of the three study periods will be less than 250 ml per visit i.e. less than the amount given when donating blood (a total amount of 1,000 ml over the entire study, which usually takes about 4 months to complete). During two of the four admissions to hospital they will receive a 48-hour infusion of intralipid (40 ml/hr of a 20% fat solution) and Heparin (250U/hr)) to raise plasma FFAs approximately 2-fold as we have previously described (8;54) whereas on the two other occasions they will receive an infusion of saline (salt water) for 48 hours in hospital. Heparin is stimulates an important enzyme involved in the breakdown of fat particles (lipoprotein lipase) and is used for this purpose in this study. Intralipid is a fat emulsions that supplies the synthetic triglycerides as substrate for LPL in order to raise plasma FFAs. Subjects will be permitted to eat and drink and will be provided with regular low fat meals during the 48 hours of the study.

ELIGIBILITY:
Inclusion Criteria:

Body mass index (BMI) > 27kg/m2. Fasting triglycerides > 2 mmol/l and < 5mmol/l Waist circumference > 90 cm Fasting blood glucose < 7 mmol/l Hemoglobin above 130g/L.

Exclusion Criteria:

* History of hepatitis/hepatic disease that has been active within the previous two years
* any significant aactive disease of the gastrointestinal, pulmonary, neurological, renal, genitourinary,hematological systems or has severe uncontrolled treated or untreated hypertension or proliferative retinopathy
* fasting blood glucose > 7mmol/l or known diabetes
* History of MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or hkeart failure
* any laboratory values>2x the upper limit of normal
* known or suspected allergy to the mediction or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions, History of hypersensitivity to heparin
* current addiction to alcohol or substances of abuse as determined by the investigator
* Metal incapacity, unwillingness or language barrier precdluding adequate understanding or cooperation
* any lipid lowering or hypoglycemic agents
* previous history of asthma
* will not donate blood thre months prior to and three months post study procedures thrombocytopenis

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
we will measure insulin secretion, calculate disposition index and insulin clearance during a hyperglycemic clamp. We will also measure insulin sensitivity during a euglycemic hyperinsulinemic clamp | one year

SECONDARY OUTCOMES:
During the hyperglycemic clamp we will also measure Free Fatty Acid, C-peptide and triyglycerides. During the euglycemic hyperinsulinemic clamp we will determine the insulin sensitivity index and the disposition index. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary F. Lewis, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada